CLINICAL TRIAL: NCT00956527
Title: Martial Arts as Early Intervention for Teen Drug Abuse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05-0681; R01DA018679 (NIH)
Record Dates: First submitted 2009-08-10; First posted 2009-08-11 (Estimated); Last update posted 2013-06-20 (Estimated); Status verified 2013-06

CONDITIONS: Adolescent; Substance Use
Keywords: Adolescent; Substance Use; Early Intervention; Martial Arts; Karate
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Modified traditional martial arts training (Experimental): Twice weekly hour-long training sessions. Classes will not vary significantly from those classes already taught at the karate school, with the following exceptions: 1) the focus of training will be primarily on the non-combative components of martial arts training, 2) there will be a higher instructor to student ratio, 3) belt advancement will be based not only on mastery of karate techniques, but also on achieving the predetermined goals as described above, and 4) weekly 5-10 minute talks will be delivered by the primary instructor and will consist of concepts relevant to substance abuse treatment (including both issues directly relating to drug use and the common skills deficits seen in "at risk" youth) and how these issues relate to martial arts concepts.
  Interventions: Behavioral: Modified traditional martial arts training

INTERVENTIONS:
Behavioral: Modified traditional martial arts training — Twice weekly hour-long training sessions. Classes will not vary significantly from those classes already taught at the karate school, with the following exceptions: 1) the focus of training will be primarily on the non-combative components of martial arts training, 2) there will be a higher instructor to student ratio, 3) belt advancement will be based not only on mastery of karate techniques, but also on achieving the predetermined goals as described above, and 4) weekly 5-10 minute talks will be delivered by the primary instructor and will consist of concepts relevant to substance abuse treatment (including both issues directly relating to drug use and the common skills deficits seen in "at risk" youth) and how these issues relate to martial arts concepts.

SUMMARY:
This is a Stage 1A/1B behavioral therapy development project with the aim of developing and piloting an early intervention based upon traditional martial arts for adolescents who are in the early stages of substance use/misuse.

The primary aims of this study are:

1) To develop a manualized version of an existing, typical traditional martial arts program, modified to target a reduction in substance use and the associated behavioral and psychosocial problems for adolescents in the early stages of substance use or misuse, based on principles derived from empirically-based prevention programs. 2) To obtain preliminary pilot data on recruitment feasibility, validity of assessments, and estimates of the effect size of the intervention in reducing substance use and improving prosocial behavioral and psychosocial outcomes. 3) To refine and further develop the manualized program based on pilot data and utilizing feedback from the initial cohort of participants, traditional martial arts program instructors and substance abuse treatment experts. The goals of these revisions would be to maximize the impact of the program on substance use and behavioral outcomes, while retaining the core features of a traditional martial arts program to ensure the feasibility of implementing, sustaining, and disseminating such a program in existing community-based martial arts programs. 4) To develop procedures for training interventionists (i.e., martial arts instructors and research assistants) and for monitoring program adherence to ensure fidelity. 5) To conduct a small pilot study of the refined manualized program to enable us to estimate the effect size of the intervention and provide information for estimating power for a larger randomized controlled trial should the results of this intervention prove promising in terms of positive impact on the primary and secondary outcome measures: decreased drug use and improvement in psychosocial functioning and behavioral problems (including aggression).

ELIGIBILITY:
Inclusion Criteria:

Subjects must: 1) be 13 through 17 years old, 2) be of estimated average intelligence (IQ>80), 3) have current or recent drug/alcohol use as evidenced by a history of substance use of at least 2 times in the 12 weeks prior to study inclusion, and 4) be medically healthy.

Exclusion Criteria:

Subjects will be excluded if they 1) meet criteria for substance dependence (other than for nicotine) based on consensus between the Composite International Diagnostic Interview- Substance Abuse Model (CIDI-SAM) and clinical interview, 2) have a history of or currently have psychosis (not explained by drug use), or bipolar disorder that is currently unstable, 3) are currently receiving psychotherapy or some form of behavioral therapy, 4) have a chronic medical illness or condition that would keep them from fully participating in physical activity, 5) have been started on a psychotropic medication in the 30 days prior to study inclusion, or 6) are pregnant.

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 31 (Actual)
Dates: Start 2006-05; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Change in substance use | end of trial

SECONDARY OUTCOMES:
Change in psychosocial functioning and behavioral problems | end of trial

CONTACTS AND LOCATIONS:
Overall Officials: Robert Davies, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Denver, Aurora, Colorado, United States